CLINICAL TRIAL: NCT01336244
Title: Double Blind Placebo Controlled Dose Ranging Study for the Assessment of Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Ascending Oral Doses of GLPG0778 in Healthy Male Subjects
Brief Title: GLPG0778: Multiple Ascending Oral Doses, Pharmacokinetic, Safety, and Pharmacodynamic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: GLPG0778-CL-102; 2011-000892-16 (EudraCT Number)
Record Dates: First submitted 2011-04-13; First posted 2011-04-15 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLPG0778 ascending doses (Experimental): Multiple ascending doses for 13 days, ranging from 50 mg twice daily upto a maximum to be determined during escalation.
  Interventions: Drug: GLPG0778
- Placebo (Placebo Comparator): Twice daily for 13 days, matching the scheme of the multiple ascending dose.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: GLPG0778 — capsules containing 50 or 100 mg of GLPG0778
  Arms: GLPG0778 ascending doses
Drug: placebo — multiple dose, aqueous formulation, 13 days days, matching ascending dose schedule
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of multiple ascending oral doses (MAD) of GLPG0778 given to healthy subjects for 13 days compared to placebo, and to evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of GLPG0778 after multiple oral administrations.

ELIGIBILITY:
Inclusion Criteria:

* healthy male, age 18-50 years
* body mass index (BMI) between 18-30 kg/m², inclusive.

Exclusion Criteria:

* significantly abnormal platelet function or coagulopathy
* smoking
* drug or alcohol abuse
* hypersensitivity to any of the test substances

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | Daily during treatment, up to 10 days postdose
  At every study visit, subjects will be asked whether any adverse events have occurred since start of treatment.
Evaluation of hematological, biochemical and cardiovascular parameters. | until 10 days postdose.
  On predefined timepoints during the study blood and urine samples will be taken, and cardiovascular tests (ECG, blood pressure, heart rate) recorded to assess whether the test compound causes any deviation.

SECONDARY OUTCOMES:
Pharmacokinetics of repeated doses | 24 hours postdose
  Bloodsamples are taken on various timepoints to assess how much of the study drug is taken up in the blood (absorption), how long it stays in the blood (excretion), and whether any "breakdown"-products of the drug are present (metabolism).
Pharmacodynamics (PD) of GLPG0778 | up to 10 days postdose
  To explore biomarkers of GLPG0778 activity after repeated oral administrations.

CONTACTS AND LOCATIONS:
Overall Officials: Gerben van 't Klooster, PhD, Study Director — Galapagos NV; Lien Gheyle, MD, Principal Investigator — SGS Stuivenberg
Locations (1):
- SGS Stuivenberg, Antwerp, Belgium